CLINICAL TRIAL: NCT01143597
Title: Improving Hand and Arm Function After SCI
Brief Title: Improving Hand and Arm Function After Spinal Cord Injury (SCI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Edelle Field-Fote, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01HD053854 (NIH)
Record Dates: First submitted 2010-06-11; First posted 2010-06-14 (Estimated); Last update posted 2013-10-10 (Estimated); Status verified 2013-10

CONDITIONS: Spinal Cord Injury
Keywords: task-specific training; arm and hand function; corticomotor plasticity; individuals with motor-incomplete spinal cord injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Somatosensory stimulation (SS) (Active Comparator): Participants in the SS group receive median nerve electrical stimulation applied to the skin of the wrists.
  Interventions: Other: Arm and hand training
- Massed practice + somatosensory stimulation (MP+SS) (Active Comparator): Participants in the MP+SS group receive a combined intervention consisting of SS and a skill-based exercise protocol
  Interventions: Other: Arm and hand training
- Conventional resistance training (CRT) (Active Comparator): Participants in the CRT group will participate in a weight-based exercise program
  Interventions: Other: Arm and hand training

INTERVENTIONS:
Other: Arm and hand training — Individuals will receive either: somatosensory stimulation isolated or combined with a skill-based exercise protocol, or a conventional strengthening program.

SUMMARY:
The long-term goal of this project is to develop rehabilitation strategies that facilitate optimal restoration of skilled hand use in individuals with spinal cord injury (SCI). The objective of the studies proposed in this application is to determine whether a protocol of massed practice + somatosensory stimulation (MP+SS) is more effective for improving skilled hand use compared to a somatosensory stimulation (SS) alone, and to determine whether these approaches are each more effective than traditional therapy (consisting of conventional resistance training; CRT).

Specific Aim I: In individuals with chronic incomplete tetraplegia, quantify changes in skilled hand use and sensory function associated with either: massed practice training combined with somatosensory stimulation (MP+SS), somatosensory stimulation (SS), or control (conventional resistance training [CRT]), and compare differences among groups. The investigators hypothesize that:

H1.1: At the end of 4 weeks, gains in scores on standardized tests of skilled hand motor function (Jebsen-Taylor Hand Function Test and Chedoke-McMaster Arm and Hand Activity Inventory) and sensory function (quantitative sensory tests; QST) will be greater in individuals who are trained using MP+SS compared to the SS and RT groups.

H1.2: At the end of 4 weeks, gains in scores on standardized tests of skilled hand motor function and sensory function tests will be greater in individuals who are trained using SS compared to CRT.

H1.3: At 6 months post training, motor and sensory gains will be retained by the MP+SS and SS groups.

Specific Aim 2: In individuals with chronic incomplete tetraplegia, quantify changes in cortical and spinal neurophysiology associated with either: massed practice combined with somatosensory stimulation (MP+SS), somatosensory stimulation (SS), or control (conventional resistance training [CRT]), and compare differences among groups. The investigators hypothesize that, after 4 weeks:

H2.1: Measures representing cortical neurophysiologic function (i.e., motor-evoked potential amplitude and location of cortical map) will show greater change in the direction of more normal values in individuals who are trained using MP+SS compared to the SS and the CRT groups.

H2.2: Measures representing spinal neurophysiologic function (i.e., F-wave and H-reflex amplitude) will show greater change in the direction of more normal values in individuals who are trained using SS compared to the MP+SS and the CRT groups.

H2.3: There will be a positive relationship between change scores associated with functional outcome measures and cortical neurophysiologic outcome measures in the MP+SS group; there will be a positive relationship between change scores associated with the functional outcome measures and spinal neurophysiologic outcome measures in the SS group.

Specific Aim 3: In individuals with chronic incomplete tetraplegia, quantify changes in self-assessment of quality of life and societal participation associated with massed practice combined with somatosensory stimulation (MP+SS), somatosensory stimulation (SS) or control (conventional resistance training [CRT]), and compare difference among groups. The investigators hypothesize that:

H3.1: Gains in scores on standardized measures of quality of life (Medical Outcomes Study Short Form 36 [SF-36]) and societal participation (Impact on Participation and Autonomy Questionnaire [IPAQ]) will be greater in individuals who are trained using MP+SS compared to both the SS and the CRT groups.

H3.2: Gains in scores on standardized measures of quality of life and societal participation will be greater in individuals who are trained using SS compared to the CRT group.

H3.3: At 6 months post training, gains in the quality of life and the societal participation measures will be retained by the MP+SS and SS groups.

Risks: This is a low risk study that investigates the effects of standard rehabilitation and exercise interventions on hand/arm function in individuals with SCI. All devices are considered minimal risk devices by the FDA.

DETAILED DESCRIPTION:
Evidence suggests that both intensive, skill-based practice training combined with somatosensory stimulation (MP+SS) and somatosensory stimulation alone (SS) may be associated with functional changes that are greater than those associated with skill-based training alone (MP). These studies are significant in that they advance the field of rehabilitation science as it relates to the goal of improving skilled hand use in individuals with SCI; there are few goals that have more important implications for function, independence and quality of life in these individuals.

ELIGIBILITY:
Inclusion Criteria:

* traumatic spinal cord injury of at least one-year duration
* injury to cervical spinal cord at C7 or higher
* sufficient strength of thenar muscles to generate, at minimum, a visible twitch contraction in at least one thumb

Exclusion Criteria:

* history of head trauma and/or cognitive deficit
* subject history of stroke, seizures or other intracranial disease
* family history of seizures
* inability to provide informed consent

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2007-08; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
The Jebsen-Taylor Hand Function Test | 4 weeks
  The Jebsen Test is an assessment of hand function and improvement in hand function associated with therapeutic procedures. Individuals with cervical SCI are included in the target population for use of the test. The test is comprised of 7 subtests, including writing, turning over cards, picking up small common objects, simulated feeding, stacking checkers, picking up large light objects, and picking up large heavy objects.

SECONDARY OUTCOMES:
Cortical motor excitability via transcranial magnetic stimulation (TMS) | 4 weeks
  The motor threshold (intensity required to evoke 5/10 motor evoked potentials), a recruitment curve (from 80% of the motor threshold to the maximum stimulator output, in increments of 20%), and the thenar motor map (number of active sites for the thenar muscles in the hand motor cortical distribution) will be recorded via TMS.

CONTACTS AND LOCATIONS:
Overall Officials: Edelle C Field-Fote, PT, PhD, Principal Investigator — University of Miami
Locations (1):
- The Miami Project to Cure Paralysis, Miami, Florida, United States

REFERENCES:
- [Background] Beekhuizen KS, Field-Fote EC. Sensory stimulation augments the effects of massed practice training in persons with tetraplegia. Arch Phys Med Rehabil. 2008 Apr;89(4):602-8. doi: 10.1016/j.apmr.2007.11.021. PMID 18373988
- [Background] Hoffman LR, Field-Fote EC. Cortical reorganization following bimanual training and somatosensory stimulation in cervical spinal cord injury: a case report. Phys Ther. 2007 Feb;87(2):208-23. doi: 10.2522/ptj.20050365. Epub 2007 Jan 9. PMID 17213410
- [Background] Beekhuizen KS, Field-Fote EC. Massed practice versus massed practice with stimulation: effects on upper extremity function and cortical plasticity in individuals with incomplete cervical spinal cord injury. Neurorehabil Neural Repair. 2005 Mar;19(1):33-45. doi: 10.1177/1545968305274517. PMID 15673842